CLINICAL TRIAL: NCT00046072
Title: A Double-Blind, Placebo-Controlled Study of E5564, A Lipid A Antagonist, Administered by Twice Daily Infusions in Patients With Severe Sepsis
Brief Title: A Safety and Efficacy Study of Intravenous E5564 in Patients With Severe Sepsis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: E5564-A001-201
Record Dates: First submitted 2002-09-19; First posted 2002-09-20 (Estimated); Last update posted 2005-12-12 (Estimated); Status verified 2005-12

CONDITIONS: Sepsis; Shock, Septic; Sepsis Syndrome; Septicemia; Infection
Keywords: Sepsis; Shock; Septic; Sepsis Syndrome; Septicemia; Endotoxins; Endotoxemia; Infection
MeSH Terms: conditions — Sepsis; Shock, Septic; Systemic Inflammatory Response Syndrome; Infections; Shock; Endotoxemia | interventions — E5564

INTERVENTIONS:
Drug: E5564

SUMMARY:
Sepsis is a serious condition where there is inflammation and damage to body tissue, usually caused by an infection. This infection can lead to decreased function of vital body organs and in some cases may lead to permanent health problems or death.

Much of the injury is due to endotoxin, a harmful substance produced by certain types of bacteria. An endotoxin antagonist is designed to block the effects of endotoxin.

This study is designed to study the safety and efficacy when treating patients with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Presently admitted, or about to be transferred, to the ICU.
* Women of Child-bearing potential must have a negative serum (or urine) hCG assay within 24 hours prior to drug administration.
* Any Race.
* Severe Sepsis [newly developed respiratory failure, refractory shock, renal dysfunction, hepatic dysfunction, or metabolic acidosis and at least three signs of SIRS (systematic inflammatory response syndrome)].
* Objective signs of infection likely to be caused by a bacterial or fungal pathogen.
* Patients must receive study medication within 8 to 12 hours of recognition of the initial sepsis-related organ failure.
* APACHE Predicted risk of mortality score between 20% and 80%.
* An intent by physicians and family to aggressively treat the patient for the 28 day study period.

Exclusion Criteria:

* Cardiogenic or hypovolemic shock.
* Acute third degree burns involving >20% of body surface.
* Recipients of non-autologous organ transplants within the past year.
* Pregnancy.
* Chronic vegetative state.
* Uncontrolled serious hemorrhage (.2 units of blood/platelets in the previous 24 hours). Patients may be considered for enrollment if bleeding has stopped and patients are still otherwise qualified.
* Unwilling or unable to be fully evaluated for all follow-up visits.
* Patients who are classified as "Do not resusitate" or "Do not treat."
* Patients who develop severe sepsis <36 hours post trauma or post-surgery. Patients may be considered for enrollment >36 hours post-trauma or post-surgery, if they meet other inclusion criteria.
* Patients with a predicted risk of mortality score of <20% or >80% after recognition of qualifying organ failure.
* Patients with a predicted risk of mortality of <51% for whom Xigris® use is planned.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-10; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Alec Wittek, M.D., Study Director — Eisai Inc.
Locations (17):
- United States (17):
  - Mobile, Alabama
  - San Diego, California
  - Santa Barbara, California
  - Jacksonville, Florida
  - Miami, Florida
  - Pensacola, Florida
  - Columbus, Georgia
  - Elk Grove, Illinois
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Buffalo, New York
  - Manhasset, New York
  - Oklahoma City, Oklahoma
  - Dallas, Texas
  - Galveston, Texas
  - San Antonio, Texas